CLINICAL TRIAL: NCT03737981
Title: A Randomized Phase III Study of Ibrutinib Plus Obinutuzumab Versus Ibrutinib Plus Venetoclax and Obinutuzumab in Untreated Older Patients (>/= 65 Years of Age) With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Testing the Addition of a New Anti-cancer Drug, Venetoclax, to the Usual Treatment (Ibrutinib and Obinutuzumab) in Untreated, Older Patients With Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02485; NCI-2018-02485 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A041702 (Other: Alliance for Clinical Trials in Oncology); A041702 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; obinutuzumab; Observation; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ibrutinib, obinutuzumab) (Active Comparator): Patients receive ibrutinib PO QD on days 1-28. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Treatment repeats every 28 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 15, patients receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Biological: Obinutuzumab
- Arm II (ibrutinib, obinutuzumab, venetoclax) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Beginning cycle 3, patients also receive venetoclax PO QD on days 1-28. Treatment repeats every 28 days for 14 cycles in the absence of disease progression or unacceptable toxicity. All patients will then receive a 15th cycle of ibrutinib. Beginning cycle 16, patients who do not achieve a BM MRD negative CR, receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a BM MRD negative CR undergo observation every 3 cycles for 6 years, then every 6 cycles thereafter.
  Interventions: Drug: Ibrutinib; Biological: Obinutuzumab; Other: Observation Activity; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA 101; GA-101; GA101; Gazyva; huMAB(CD20); R 7159; R-7159; R7159; RO 5072759; RO-5072759; RO5072759
Other: Observation Activity — Undergo observation
  Other Names: Observation
  Arms: Arm II (ibrutinib, obinutuzumab, venetoclax)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Arm II (ibrutinib, obinutuzumab, venetoclax)

SUMMARY:
This phase III trial compares adding a new anti-cancer drug (venetoclax) to the usual treatment (ibrutinib plus obinutuzumab) in older patients with chronic lymphocytic leukemia who have not received previous treatment. The addition of venetoclax to the usual treatment might prevent chronic lymphocytic leukemia from returning. This trial also will investigate whether patients who receive ibrutinib plus obinutuzumab plus venetoclax and have no detectable chronic lymphocytic leukemia after 1 year of treatment, can stop taking ibrutinib. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with obinutuzumab may induce changes in body's immune system and may interfere with the ability of cancer cells to grow and spread. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving ibrutinib and obinutuzumab with venetoclax may work better at treating chronic lymphocytic leukemia compared to ibrutinib and obinutuzumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the progression-free survival (PFS) between control treatment and experimental treatment strategies: ibrutinib/obinutuzumab (IO) with ibrutinib maintenance (IM) versus ibrutinib/venetoclax/obinutuzumab (IVO) regardless of IM or observation.

SECONDARY OBJECTIVES:

I. To compare bone marrow (BM) minimal residual disease (MRD)- complete response (CR) rates, MRD- rates, and depth of response at cycle 15 day 1 between patients treated with IO versus IVO.

II. To compare overall survival (OS) between the control and experimental treatment strategies: IO with IM versus IVO regardless of IM or observation.

III. To compare the 5-year PFS and overall survival (OS) for the control and experimental treatment strategies: IO with IM versus IVO regardless of IM or observation.

IV. To describe the toxicity profile for each of the treatment strategies and by each treatment course.

CORRELATIVES SCIENCE OBJECTIVES:

I. To compare MRD status between blood and bone marrow at the end of induction treatment/cycle 15 day 1 to determine whether blood MRD can be used as a surrogate to bone marrow MRD with these treatment regimens.

II. To compare peripheral blood MRD status by standard central flow cytometry to next generation sequencing (NGS) using ClonoSeq technique to determine the agreement in MRD negativity of the two techniques.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Patients also receive obinutuzumab intravenously (IV) on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Treatment repeats every 28 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 15, patients receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive ibrutinib PO QD on days 1-28. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Beginning cycle 3, patients also receive venetoclax PO QD on days 1-28. Treatment repeats every 28 days for 14 cycles in the absence of disease progression or unacceptable toxicity. All patients will then receive a 15th cycle of ibrutinib. Beginning cycle 16, patients who do not achieve a BM MRD negative CR, receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a BM MRD negative CR undergo observation every 3 cycles for 6 years, then every 6 cycles thereafter.

After completion of study treatment, patients are followed every 6 months until 10 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY CRITERIA (STEP 0)
* Patients must have been diagnosed with chronic lymphocytic leukemia (CLL) (> 5000 B-cells per uL of peripheral blood at any point during the course of their disease) or small lymphocytic lymphoma (SLL) with < 5000 B-cells per uL of blood but with disease-associated lymphadenopathy
* This blood submission is mandatory prior to registration/randomization to perform fluorescence in situ hybridization (FISH) centrally that will be used for stratification. It should be obtained as soon after pre-registration as possible
* REGISTRATION ELIGIBILITY CRITERIA (STEP 1)
* Patients must be diagnosed with CLL or SLL in accordance with 2018 International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria that includes all of the following:

  * >= 5 x10^9 B lymphocytes (5000/uL) in the peripheral blood measured by flow cytometry at any point in the course of the disease or less peripheral blood involvement but disease-associated lymphadenopathy
  * On local morphologic review, the leukemic cells must be small mature lymphocytes, and prolymphocytes must not exceed 55% of the blood lymphocytes
  * Neoplastic cells on immunophenotype (performed locally) must reveal a clonal B-cell population, which express the B cell surface markers of CD19 and CD20, as well as the T-cell antigen CD5. Patients with bright surface immunoglobulin expression or lack of CD23 expression in >10% of cells must lack t(11;14) translocation by interphase cytogenetics
* Patients must be intermediate or high-risk Rai stage CLL or SLL

  * Intermediate risk (formerly stage I/II) is defined by lymphadenopathy and/or hepatomegaly or splenomegaly without anemia or thrombocytopenia
  * High risk (formerly stage III/IV) is defined by splenomegaly and/or anemia (hemoglobin < 11g/dL) not attributable to autoimmune hemolytic anemia and/or thrombocytopenia (platelets [plt] < 100 x10^9/L) not attributable to autoimmune thrombocytopenia
* Patients must meet criteria for treatment as defined by 2018 IWCLL guidelines which includes at least one of the following criteria:

  * Evidence of marrow failure as manifested by the development or worsening of anemia or thrombocytopenia (not attributable to autoimmune hemolytic anemia or thrombocytopenia)
  * Massive (>= 6 cm below the costal margin), progressive or symptomatic splenomegaly
  * Massive nodes (>= 10 cm) or progressive or symptomatic lymphadenopathy
  * Progressive lymphocytosis with a lymphocyte doubling time < 6 months or an increase of >= 50% over a 2 month period
  * Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy
  * Symptomatic or functional extranodal involvement (e.g. skin, kidney, lung, spine)
  * Constitutional symptoms, which include any of the following:

    * Unintentional weight loss of 10% or more within 6 months
    * Significant fatigue
    * Fevers > 100.5 degrees Fahrenheit (F) for 2 weeks or more without evidence of infection
    * Night sweats >= 1 month without evidence of infection
* Treatment with rituximab and/or high dose corticosteroids for autoimmune complications of CLL/SLL must be complete at least 4 weeks prior to enrollment. Palliative steroids must be at a dose not higher than 20 mg/day of prednisone or equivalent corticosteroid at the time of registration
* Age >= 65 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,000/mm^3 except if due to bone marrow involvement
* Platelet count (untransfused) >= 30,000/mm^3 except if due to bone marrow involvement
* Calculated (Calc.) creatinine clearance >= 40 mL/min (by Cockcroft-Gault)
* Bilirubin =< 1.5 x upper limit of normal (ULN) except if due to liver involvement, hemolysis, or Gilbert's disease
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN) except if due to liver involvement
* If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated
* Please note: Intravenous immunoglobulin therapy (IVIG) can cause a false positive hepatitis B serology. If patients receiving routine IVIG have core antibody or surface antigen positivity without evidence of active viremia (negative hepatitis B deoxyribonucleic acid [DNA]) they may still participate in the study, must have hepatitis serologies and hepatitis B DNA monitored periodically by the treating physician
* If history of hepatitis C virus (HCV) infection, must be treated with undetectable HCV viral load
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Central fluorescent in situ hybridization (FISH) blood results are mandatory prior to registration/randomization for it will be used for stratification
* Patients must be able to swallow capsules and not have the following conditions: disease significantly affecting gastrointestinal absorption, resection of the stomach or small bowel, partial or complete bowel obstruction
* Patients must be able to receive either a xanthine oxidase inhibitor or rasburicase for prophylaxis/treatment of tumor lysis syndrome (TLS)
* RE-REGISTRATION ELIGIBILITY CRITERIA (STEP 2)
* Completion of treatment through cycle 14 day 28, and remain on ibrutinib therapy
* Receipt of central BM MRD results
* Response assessment completed with CR determination

Exclusion Criteria:

* Patients must not have had prior therapy for CLL/SLL (except palliative steroids or treatment of autoimmune complications of CLL with rituximab or steroids)
* Patients must not have any history of Richter's transformation or prolymphocytic leukemia (prolymphocytes in blood > 55%)
* Patients with class III or class IV heart failure by New York Heart Association, those with unstable angina, and those with uncontrolled arrhythmia are not eligible
* Patients who have had a myocardial infarction, intracranial bleed, or stroke within the past 6 months are not eligible
* Patients must not be receiving active systemic anticoagulation with heparin or warfarin. Patients on warfarin must discontinue the drug for at least 10 days prior to registration on the study
* Chronic concomitant treatment with strong inhibitors of CYP3A4/5 is not allowed on this study. Patients on strong CYP3A inhibitors must discontinue the drug for 14 days prior to registration on the study
* Chronic concomitant treatment with strong CYP3A4/5 inducers is not allowed. Patients must discontinue the drug 14 days prior to registration on the study
* Patients must not require more than 20 mg prednisone or equivalent corticosteroid daily
* Patients must not have uncontrolled active systemic infection requiring intravenous antibiotics
* Patients must not have a known allergy to mannitol
* Patients must not have prior significant hypersensitivity to rituximab (not including infusion reactions)
* Patients may not have had major surgery within 10 days prior to registration, or minor surgery within 7 days prior to registration. Examples of minor surgery include dental surgery, insertion of a venous access device, skin biopsy, or aspiration for a joint. The decision about whether a surgery is major or minor can be made at the discretion of the treating physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 465 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2026-06-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Woyach, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (860):
- United States (860):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Broward Health North, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Island Urology-Hilo, Hilo, Hawaii
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Mission Hospital, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Novant Health Cancer Institute - Statesville, Stateville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wpafb, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - STCC at DHR Health Institute for Research and Development, Edinburg, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 534 patients were pre-registered, 465 went on to register and were randomized to treatment
Groups:
- Arm I (Ibrutinib, Obinutuzumab): Patients receive ibrutinib PO QD on days 1-28. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Treatment repeats every 28 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 15, patients receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Ibrutinib: Given PO
  >
  > Obinutuzumab: Given IV
- Arm II (Ibrutinib, Obinutuzumab, Venetoclax): Patients receive ibrutinib PO QD on days 1-28. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Beginning cycle 3, patients also receive venetoclax PO QD on days 1-28. Treatment repeats every 28 days for 14 cycles in the absence of disease progression or unacceptable toxicity. All patients will then receive a 15th cycle of ibrutinib. Beginning cycle 16, patients who do not achieve a BM MRD negative CR, receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a BM MRD negative CR undergo observation every 3 cycles for 6 years, then every 6 cycles thereafter.
  >
  > Ibrutinib: Given PO
  >
  > Obinutuzumab: Given IV
  >
  > Observation Activity: Undergo observation
  >
  > Venetoclax: Given PO
Period: Initial Treatment
Arm/Group | Arm I (Ibrutinib, Obinutuzumab) | Arm II (Ibrutinib, Obinutuzumab, Venetoclax)
Started | 232 | 233
Completed | 166 | 158
Not Completed | 66 | 75
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Adverse Event | 32 | 22
Not completed — Disease progression | 1 | 4
Not completed — Alternative therapy | 1 | 1
Not completed — Complicating disease | 8 | 6
Not completed — Death | 11 | 15
Not completed — Patient withdrawal prior to treatment | 1 | 2
Not completed — Patient not on Ibrutinib | 0 | 1
Not completed — Patient moved | 0 | 1
Not completed — Patient ineligible | 0 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Death prior to treatment | 0 | 1
Not completed — Patient inability to follow protocol | 0 | 1
Not completed — Other | 4 | 9
Period: Subsequent Ibrutinib/Observation
Arm/Group | Arm I (Ibrutinib, Obinutuzumab) | Arm II (Ibrutinib, Obinutuzumab, Venetoclax)
Started | 166 | 158 (53 patients in arm II went on to subsequent Ibrutinib treatment, 105 went on to observation)
Completed | 0 | 2
Not Completed | 166 | 156
Not completed — Withdrawal by Subject | 11 | 7
Not completed — Adverse Event | 38 | 12
Not completed — Disease progression | 3 | 3
Not completed — Alternative therapy | 1 | 2
Not completed — Complicating disease | 4 | 5
Not completed — Death | 13 | 16
Not completed — Other | 2 | 7
Not completed — On treatment | 90 | 101
Not completed — Physician Decision | 3 | 1
Not completed — Clinical response | 1 | 1
Not completed — VA denial of authorization | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Ibrutinib, Obinutuzumab): Patients receive ibrutinib PO QD on days 1-28. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Treatment repeats every 28 days for up to 14 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 15, patients receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity.> > Ibrutinib: Given PO>
  > Obinutuzumab: Given IV
- Arm II (Ibrutinib, Obinutuzumab, Venetoclax): Patients receive ibrutinib PO QD on days 1-28. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1, and on day 1 of cycles 2-6. Beginning cycle 3, patients also receive venetoclax PO QD on days 1-28. Treatment repeats every 28 days for 14 cycles in the absence of disease progression or unacceptable toxicity. All patients will then receive a 15th cycle of ibrutinib. Beginning cycle 16, patients who do not achieve a BM MRD negative CR, receive ibrutinib PO QD every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a BM MRD negative CR undergo observation every 3 cycles for 6 years, then every 6 cycles thereafter.> > Ibrutinib: Given PO>
  > Obinutuzumab: Given IV>
  > Observation Activity: Undergo observation>
  > Venetoclax: Given PO
- Total: Total of all reporting groups
Arm/Group | Arm I (Ibrutinib, Obinutuzumab) | Arm II (Ibrutinib, Obinutuzumab, Venetoclax) | Total
Number analyzed (Participants) | 232 | 233 | 465
Age, Continuous [Median (Full Range); unit: years] | 74 [65 to 89] | 74 [65 to 89] | 74 [65 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 82 | 151
  Male | 163 | 151 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 218 | 223 | 441
  Unknown or Not Reported | 13 | 7 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 16 | 24
  White | 214 | 210 | 424
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 232 | 233 | 465
Rai Stage classification category [Count of Participants; unit: Participants] — Intermediate Risk (Formerly Stage I/II) - Lymphadenopathy and/or hepatomegaly or splenomegaly without anemia or thrombocytopenia>
  > High Risk (Formerly Stage III/IV) - Splenomegaly and/or Anemia (hemoglobin <11g/dL) not attributable to autoimmune hemolytic anemia and/or Thrombocytopenia (plt <100 x109/L) not attributable to autoimmune thrombocytopenia
  Participants
    High | 129 | 129 | 258
    Intermediate | 103 | 104 | 207
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction>
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work>
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours>
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours>
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair>
  5. Dead
  Participants
    0 | 119 | 114 | 233
    1 | 106 | 111 | 217
    2 | 7 | 8 | 15
High-risk FISH abnormality del(17p13.1) [Count of Participants; unit: Participants] — Deletion on the short arm of chromosome 17 determined by fluorescence in Situ Hybridization (FISH) is present or absent
  Participants
    Absent | 202 | 202 | 404
    Present | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS will be compared between the experimental and control treatment strategy groups using a stratified log-rank test (stratified on Rai stage, intermediate versus [vs.] high, and del(17p13.1) by fluorescence in situ hybridization [FISH], present vs. absent). The Kaplan-Meier method will be used to estimate PFS distributions. Five-year PFS estimates and corresponding hazard ratios will be provided with 95% confidence intervals for each treatment strategy.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants w/out event
Arm/Group | Arm I (Ibrutinib, Obinutuzumab) | Arm II (Ibrutinib, Obinutuzumab, Venetoclax)
Number analyzed (Participants) | 232 | 233
proportion of participants w/out event | 0.59 [0.51 to 0.67] | 0.68 [0.61 to 0.75]
Statistical Analysis 1: Comparison: Arm I (Ibrutinib, Obinutuzumab) vs Arm II (Ibrutinib, Obinutuzumab, Venetoclax); Test type: Superiority; p = 0.2414, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.64 to 1.24]

2. Secondary Outcome: Bone Marrow (BM) Minimal Residual Disease (MRD)- Complete Response (CR) Rate
Description: BM MRD- CR rate will be calculated and will be estimated using the number of patients meeting the BM MRD- CR criteria divided by the total number of patients randomized to each of the treatment arms. The stratified Cochran-Mantel-Haenszel test will be used to compare the BM MRD- CR rates between treatment arms (stratified on Rai stage, intermediate vs. high, and del(17p13.1) by FISH, present vs. absent).
Time Frame: Up to 10 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate the OS distribution for each treatment strategy. Estimates at 5 years will be calculated with corresponding 95% confidence intervals, and differences in these estimates between the treatment strategies will be tested using a stratified chi-square test based on the complementary log-log transformation of the Kaplan-Meier estimates. Comparisons in OS curves between experimental and control treatment strategies will use a stratified log-rank test (stratified on Rai stage, intermediate vs. high, and del(17p13.1) by FISH, present vs. absent). Hazard ratios with 95% confidence intervals will be estimated from the corresponding, stratified proportional hazard model.
Time Frame: From randomization date until death from any cause, assessed up to 10 years
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Adverse Events
Description: Will be defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment, graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Frequency and severity of adverse events and tolerability for each treatment strategy group will be summarized using descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. The incidence of severe (grade 3+) adverse events or toxicities will be described.
Time Frame: Up to 10 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6.75 years
Groups:
- Arm I (Ibrutinib, Obinutuzumab): Ibrutinib 420 mg PO daily days 1-28 for 15 cycles Obinutuzumab 100 mg IV 100 mg on C1D1, 900 mg on C1D2, 1000 mg on Cycle1D8 & C1D15, C2-6D1
- Arm II (Ibrutinib, Obinutuzumab, Venetoclax): Ibrutinib 420 mg PO daily days 1-28 for 15 cycles Obinutuzumab 100 mg IV 100 mg on C1D1, 900 mg on C1D2, 1000 mg on C1D8 & C1D15, C2-6D1 Venetoclax 20 mg daily PO beginning C3D1, dose escalated weekly to a final dose of 400 mg on C4D1, then 400 mg daily PO C4D1-C14D28
- Subsequent Treatment - Ibrutinib: Ibrutinib 420 mg PO daily days 1-28 until progression or unacceptable adverse events
- Subsequent Treatment - Observation: q3 cycles for 6 years from registration, then q6 cycles until progression
Arm/Group | Arm I (Ibrutinib, Obinutuzumab) | Arm II (Ibrutinib, Obinutuzumab, Venetoclax) | Subsequent Treatment - Ibrutinib | Subsequent Treatment - Observation
All-Cause Mortality (participants affected / at risk) | 11/232 | 15/233 | 20/219 | 9/105
Serious Adverse Events (participants affected / at risk) | 0/232 | 0/233 | 0/219 | 0/105
Other Adverse Events (participants affected / at risk) | 229/232 | 230/233 | 213/219 | 104/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Ibrutinib, Obinutuzumab) (N=232) | Arm II (Ibrutinib, Obinutuzumab, Venetoclax) (N=233) | Subsequent Treatment - Ibrutinib (N=219) | Subsequent Treatment - Observation (N=105)
Anemia (Blood and lymphatic system disorders) | 73 (197) | 87 (241) | 70 (217) | 29 (99)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 8 (40) | 5 (29) | 12 (79) | 7 (29)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 3 (5) | 1 (1) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 7 (9) | 2 (3) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 16 (23) | 18 (19) | 1 (1) | 0 (0)
Methemoglobinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 42 (131) | 53 (184) | 68 (298) | 18 (76)
Atrial flutter (Cardiac disorders) | 4 (11) | 3 (3) | 4 (9) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (16)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (5) | 1 (1) | 9 (46) | 6 (44)
Chest pain - cardiac (Cardiac disorders) | 7 (7) | 4 (5) | 3 (3) | 2 (5)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 5 (7) | 8 (9) | 5 (10) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (13)
Myocardial infarction (Cardiac disorders) | 3 (3) | 4 (4) | 7 (7) | 0 (0)
Palpitations (Cardiac disorders) | 18 (37) | 10 (15) | 3 (10) | 3 (3)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (16)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 10 (11) | 9 (26) | 18 (82) | 8 (25)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 7 (8) | 5 (5) | 2 (3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (16)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Congen, family, genetic disord -Oth spec (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 5 (5) | 2 (4) | 2 (15) | 5 (8)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 4 (8) | 5 (16) | 7 (51) | 4 (26)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 4 (18) | 3 (11) | 2 (10) | 2 (5)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 5 (13) | 2 (3) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 1 (1) | 3 (5) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 1 (2) | 0 (0) | 1 (11) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (3) | 0 (0) | 4 (21) | 3 (6)
Testosterone deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (9)
Blurred vision (Eye disorders) | 7 (13) | 6 (11) | 7 (29) | 1 (1)
Cataract (Eye disorders) | 3 (6) | 0 (0) | 4 (16) | 3 (17)
Dry eye (Eye disorders) | 2 (9) | 5 (14) | 4 (12) | 1 (11)
Eye disorders - Other, specify (Eye disorders) | 6 (13) | 10 (25) | 11 (24) | 2 (2)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (3) | 1 (3) | 1 (6)
Glaucoma (Eye disorders) | 1 (2) | 0 (0) | 1 (6) | 1 (12)
Periorbital edema (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (4) | 1 (3) | 0 (0) | 1 (9)
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (3) | 0 (0) | 2 (5) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (18) | 14 (35) | 14 (26) | 6 (14)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Belching (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 6 (11) | 5 (8) | 3 (5) | 2 (3)
Cheilitis (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 27 (59) | 25 (60) | 20 (40) | 16 (68)
Dental caries (Gastrointestinal disorders) | 2 (3) | 1 (2) | 0 (0) | 1 (15)
Diarrhea (Gastrointestinal disorders) | 87 (242) | 159 (559) | 88 (381) | 35 (103)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 11 (27) | 7 (15) | 3 (19)
Dyspepsia (Gastrointestinal disorders) | 7 (23) | 20 (55) | 11 (25) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 6 (6) | 6 (12) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (2) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (6) | 10 (16) | 3 (8) | 2 (16)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (17) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 14 (48) | 10 (41) | 12 (45) | 5 (22)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 8 (17) | 17 (28) | 12 (33) | 4 (17)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 4 (10) | 0 (0) | 4 (5) | 1 (15)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 20 (42) | 25 (50) | 13 (49) | 0 (0)
Nausea (Gastrointestinal disorders) | 41 (83) | 65 (165) | 19 (35) | 8 (38)
Oral dysesthesia (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (7) | 3 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 6 (9) | 4 (7) | 4 (17) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3) | 2 (10)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (15) | 29 (49) | 14 (19) | 3 (3)
Chills (General disorders and administration site conditions) | 19 (23) | 24 (33) | 4 (5) | 1 (1)
Death NOS (General disorders and administration site conditions) | 0 (0) | 4 (4) | 3 (3) | 1 (1)
Edema face (General disorders and administration site conditions) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Edema limbs (General disorders and administration site conditions) | 87 (329) | 82 (331) | 102 (644) | 22 (91)
Facial pain (General disorders and administration site conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders and administration site conditions) | 175 (933) | 185 (1004) | 157 (1162) | 74 (386)
Fever (General disorders and administration site conditions) | 20 (21) | 23 (24) | 13 (13) | 2 (2)
Flu like symptoms (General disorders and administration site conditions) | 7 (10) | 5 (6) | 4 (4) | 2 (2)
Gait disturbance (General disorders and administration site conditions) | 5 (9) | 1 (4) | 8 (27) | 2 (2)
Gen disord and admin site conds-Oth spec (General disorders and administration site conditions) | 14 (30) | 9 (18) | 6 (14) | 3 (8)
Generalized edema (General disorders and administration site conditions) | 0 (0) | 2 (3) | 1 (1) | 1 (4)
Hypothermia (General disorders and administration site conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infusion site extravasation (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders and administration site conditions) | 3 (7) | 1 (1) | 2 (7) | 1 (1)
Malaise (General disorders and administration site conditions) | 5 (15) | 3 (4) | 2 (8) | 0 (0)
Multi-organ failure (General disorders and administration site conditions) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Neck edema (General disorders and administration site conditions) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders and administration site conditions) | 6 (13) | 8 (9) | 6 (6) | 2 (6)
Pain (General disorders and administration site conditions) | 16 (25) | 11 (22) | 12 (30) | 9 (20)
Sudden death NOS (General disorders and administration site conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (7) | 2 (2) | 0 (0)
Gallbladder fistula (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (4)
Allergic reaction (Immune system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (5)
Immune system disorders - Other, specify (Immune system disorders) | 3 (4) | 1 (2) | 6 (32) | 3 (8)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 3 (3)
Bone infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (5) | 1 (3) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 5 (7) | 3 (3) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (7) | 1 (1)
Folliculitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (4) | 0 (0)
Fungemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gum infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Herpes simplex reactivation (Infections and infestations) | 4 (9) | 2 (6) | 0 (0) | 1 (6)
Infections and infestations - Oth spec (Infections and infestations) | 28 (40) | 43 (55) | 68 (93) | 21 (43)
Joint infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 21 (25) | 28 (37) | 47 (76) | 11 (16)
Nail infection (Infections and infestations) | 4 (4) | 1 (2) | 5 (7) | 1 (4)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Otitis media (Infections and infestations) | 1 (2) | 3 (5) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (2) | 2 (7) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 5 (10) | 1 (2)
Penile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 13 (14) | 8 (8) | 2 (2)
Shingles (Infections and infestations) | 3 (4) | 4 (4) | 3 (5) | 1 (1)
Sinusitis (Infections and infestations) | 7 (15) | 4 (7) | 13 (29) | 4 (20)
Skin infection (Infections and infestations) | 8 (13) | 12 (18) | 19 (32) | 4 (5)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 4 (6) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 10 (15) | 9 (15) | 18 (29) | 9 (15)
Urinary tract infection (Infections and infestations) | 22 (33) | 16 (26) | 24 (32) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Viremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 3 (4) | 4 (5) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 137 (612) | 143 (673) | 135 (997) | 45 (181)
Burn (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 12 (16) | 16 (18) | 22 (30) | 6 (7)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (9) | 10 (13) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 32 (34) | 31 (34) | 0 (0) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 3 (3) | 3 (5) | 6 (9) | 4 (16)
Injury to jugular vein (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 1 (3) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Urethral anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Activated partial throm time prolonged (Investigations) | 2 (2) | 3 (3) | 1 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 12 (20) | 26 (40) | 18 (33) | 3 (11)
Alkaline phosphatase increased (Investigations) | 14 (19) | 21 (47) | 18 (40) | 4 (20)
Aspartate aminotransferase increased (Investigations) | 23 (36) | 28 (45) | 20 (55) | 4 (6)
Blood bilirubin increased (Investigations) | 27 (59) | 37 (87) | 27 (96) | 13 (46)
Blood lactate dehydrogenase increased (Investigations) | 30 (60) | 35 (68) | 21 (70) | 7 (16)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (8)
Cardiac troponin I increased (Investigations) | 3 (3) | 3 (3) | 4 (4) | 0 (0)
Cardiac troponin T increased (Investigations) | 2 (2) | 2 (2) | 4 (5) | 0 (0)
Cholesterol high (Investigations) | 2 (3) | 0 (0) | 2 (5) | 4 (10)
Creatinine increased (Investigations) | 41 (107) | 42 (109) | 59 (248) | 18 (69)
ECG QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (13)
Ejection fraction decreased (Investigations) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Hemoglobin increased (Investigations) | 3 (6) | 1 (3) | 1 (5) | 1 (1)
INR increased (Investigations) | 5 (11) | 8 (18) | 7 (26) | 0 (0)
Investigations - Other, specify (Investigations) | 4 (18) | 9 (15) | 14 (71) | 11 (57)
Lipase increased (Investigations) | 1 (1) | 2 (8) | 4 (16) | 1 (3)
Lymphocyte count decreased (Investigations) | 41 (107) | 85 (284) | 61 (233) | 35 (133)
Lymphocyte count increased (Investigations) | 50 (123) | 48 (81) | 14 (35) | 0 (0)
Neutrophil count decreased (Investigations) | 115 (290) | 155 (510) | 46 (117) | 23 (64)
Platelet count decreased (Investigations) | 163 (639) | 179 (872) | 102 (677) | 41 (168)
Serum amylase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 3 (4) | 2 (2) | 2 (2) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Investigations) | 8 (22) | 7 (19) | 11 (62) | 5 (23)
Weight loss (Investigations) | 10 (23) | 18 (36) | 17 (43) | 9 (29)
White blood cell decreased (Investigations) | 31 (71) | 93 (277) | 29 (69) | 17 (54)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 15 (21) | 33 (62) | 14 (18) | 3 (9)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (10) | 8 (10) | 4 (5) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 2 (6) | 1 (1) | 2 (5) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 4 (8) | 3 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 47 (126) | 45 (103) | 51 (175) | 25 (82)
Hyperkalemia (Metabolism and nutrition disorders) | 20 (36) | 16 (18) | 17 (34) | 5 (7)
Hyperlipidemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 2 (2) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 5 (11) | 11 (16) | 7 (9) | 5 (9)
Hyperphosphatemia (Metabolism and nutrition disorders) | 11 (21) | 24 (43) | 3 (5) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (7) | 0 (0) | 2 (15) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 15 (22) | 12 (15) | 10 (27) | 3 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 31 (54) | 33 (76) | 31 (68) | 5 (14)
Hypocalcemia (Metabolism and nutrition disorders) | 23 (40) | 37 (61) | 25 (49) | 6 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 16 (26) | 10 (18) | 8 (13) | 4 (10)
Hypokalemia (Metabolism and nutrition disorders) | 11 (26) | 29 (63) | 16 (23) | 5 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (11) | 12 (36) | 7 (30) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 30 (64) | 39 (75) | 30 (67) | 7 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6) | 18 (24) | 6 (12) | 2 (6)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 2 (5) | 4 (13) | 5 (6) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (8) | 1 (19) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 4 (4) | 11 (11) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 90 (358) | 109 (510) | 97 (578) | 36 (278)
Arthritis (Musculoskeletal and connective tissue disorders) | 13 (37) | 5 (12) | 11 (55) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (61) | 30 (66) | 26 (78) | 11 (51)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (16) | 4 (7) | 2 (14) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (3) | 2 (5) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 15 (28) | 18 (28) | 14 (33) | 2 (5)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 4 (5) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 39 (93) | 20 (48) | 23 (72) | 2 (9)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (7) | 3 (5) | 1 (9)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 18 (54) | 11 (33) | 18 (47) | 8 (58)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (17) | 21 (50) | 8 (20) | 7 (19)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (10) | 7 (15) | 2 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 2 (6) | 3 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (44) | 11 (16) | 29 (109) | 4 (10)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (27) | 17 (35) | 29 (63) | 13 (36)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (8) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 1 (7) | 1 (4) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (3) | 0 (0) | 3 (12) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 3 (7) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 30 (60) | 35 (67) | 15 (38) | 7 (10)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Dysesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (21) | 18 (47) | 5 (11) | 4 (6)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 2 (4) | 3 (6) | 0 (0)
Headache (Nervous system disorders) | 30 (81) | 33 (74) | 16 (48) | 5 (15)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 1 (4) | 3 (3) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 5 (15) | 2 (24) | 3 (7)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 3 (4) | 4 (4) | 6 (11) | 2 (3)
Neuralgia (Nervous system disorders) | 1 (4) | 2 (4) | 1 (1) | 1 (5)
Paresthesia (Nervous system disorders) | 6 (8) | 12 (28) | 3 (11) | 4 (16)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (6) | 3 (15) | 1 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (49) | 16 (34) | 21 (101) | 4 (12)
Presyncope (Nervous system disorders) | 1 (1) | 2 (4) | 3 (3) | 0 (0)
Reversbl posterior leukoenceph syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (3)
Somnolence (Nervous system disorders) | 4 (10) | 0 (0) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 12 (14) | 4 (4) | 3 (3)
Transient ischemic attacks (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 6 (26) | 4 (13) | 7 (45) | 1 (17)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 10 (41) | 13 (28) | 13 (90) | 4 (16)
Confusion (Psychiatric disorders) | 6 (6) | 6 (8) | 6 (6) | 1 (2)
Delayed orgasm (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 10 (21) | 2 (4) | 13 (60) | 2 (14)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 25 (47) | 18 (35) | 11 (38) | 7 (41)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 5 (6) | 13 (14) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (3)
Chronic kidney disease (Renal and urinary disorders) | 9 (22) | 8 (26) | 22 (92) | 8 (45)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (2) | 3 (7) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (3) | 2 (6) | 6 (10) | 1 (1)
Glucosuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 14 (22) | 9 (18) | 16 (34) | 7 (8)
Proteinuria (Renal and urinary disorders) | 2 (2) | 4 (5) | 4 (4) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 7 (14) | 2 (2) | 8 (10) | 0 (0)
Renal calculi (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (4) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 6 (15) | 8 (12) | 9 (20) | 3 (7)
Urinary incontinence (Renal and urinary disorders) | 4 (5) | 1 (1) | 2 (7) | 3 (5)
Urinary retention (Renal and urinary disorders) | 3 (4) | 2 (4) | 6 (28) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (4) | 4 (6) | 0 (0) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (8) | 1 (1) | 3 (29)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 3 (5) | 3 (25)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (10) | 4 (13) | 4 (12) | 3 (11)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (51) | 41 (90) | 42 (95) | 15 (54)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 40 (83) | 42 (82) | 32 (85) | 10 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 14 (25) | 10 (17) | 2 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 1 (3) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (8) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 10 (14) | 12 (13) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 10 (15) | 14 (29) | 7 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (14) | 5 (12) | 8 (12) | 0 (0)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 3 (3) | 3 (5) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4) | 8 (9) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 5 (7) | 8 (22) | 3 (5)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (9) | 0 (0) | 1 (6) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 13 (16) | 10 (34) | 7 (21)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 9 (9) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 3 (3) | 10 (30) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (10) | 4 (27) | 5 (24)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 10 (11) | 3 (8) | 3 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (8) | 2 (2) | 1 (14) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (32) | 5 (16) | 4 (11) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 19 (46) | 16 (43) | 17 (105) | 5 (42)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (12) | 7 (29) | 2 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (20) | 11 (13) | 4 (4) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (4) | 2 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 9 (26) | 6 (23) | 21 (99) | 4 (23)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 3 (5) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (35) | 19 (32) | 9 (27) | 1 (6)
Purpura (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (7) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (17) | 5 (7) | 1 (6) | 4 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 65 (159) | 70 (157) | 44 (142) | 19 (54)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 33 (68) | 20 (40) | 36 (115) | 9 (52)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 5 (6) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 5 (8) | 4 (6) | 9 (11) | 3 (4)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (3) | 5 (5) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 6 (7) | 3 (3) | 3 (3) | 1 (3)
Hot flashes (Vascular disorders) | 4 (7) | 2 (5) | 6 (14) | 3 (9)
Hypertension (Vascular disorders) | 156 (900) | 171 (947) | 158 (1368) | 81 (644)
Hypotension (Vascular disorders) | 11 (11) | 17 (17) | 9 (12) | 3 (4)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 3 (4) | 6 (14) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 2 (7) | 1 (6) | 2 (2) | 1 (13)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03737981/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03737981/ICF_001.pdf